CLINICAL TRIAL: NCT05911412
Title: Development of the Neuroimaging Biomarker-based Prediction Model of Anxiety-related Disorders and Novel Treatment Strategies: Effect of Mindfulness-based Cognitive Therapy Using Neuroscience on the Brain
Brief Title: Development of the Neuroimaging Biomarker-based Prediction Model of Anxiety-related Disorders: Effect of Mindfulness-based Cognitive Therapy Using Neuroscience on the Brain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CHA University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Sang-Hyuk Lee, Professor at Bundang CHA medical center, CHA University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-10-041-002
Record Dates: First submitted 2023-02-23; First posted 2023-06-22 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Anxiety Depression
Keywords: mindfulness-based cognitive therapy; mri; neuroscience

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMBCT intervention (Experimental): Participants in this arm enter the 8-week NMBCT course immediately after the baseline visit.
  Interventions: Behavioral: Mindfulness-based cognitive therapy using neuroscience (NMBCT)
- Waitlist (Experimental): Participants in the waitlist control arm will wait for 8 weeks after the baseline visit, and then will be offered an identical 8-week NMBCT course.
  Interventions: Behavioral: Mindfulness-based cognitive therapy using neuroscience (NMBCT)

INTERVENTIONS:
Behavioral: Mindfulness-based cognitive therapy using neuroscience (NMBCT) — Mindfulness-based cognitive therapy using neuroscience (NMBCT) is a standardized 8-week course taught by trained instructors. The NMBCT is a group therapy that takes place once a week for about 90 minutes per session. The program consists of mental education for each session, 2-3 mindfulness meditation practice, mindfulness practice in daily life, and about 30 minutes of daily home mindfulness meditation task. While participating in the program, the subjects will receive psychoeducation and various mindfulness meditation techniques (eating meditation, breathing meditation, sedentary meditation, viewing meditation, and listening meditation, etc.).

SUMMARY:
The purpose of this study designed a randomized clinical trial is to determine the efficacy of an 8-week mindfulness-based cognitive therapy using neuroscience (NMBCT) to reduce anxiety or depressive symptoms among adult participants with anxiety and depression. The primary object is to assess the effectiveness of NMBCT to change in the structural or functional brain. A secondary objective is to reduce clinical symptom severity.

DETAILED DESCRIPTION:
There are reports that mindfulness-based cognitive therapy (MBCT) techniques in patients with panic disorder or depression promote neuroplasticity changes in the brain, thereby restoring individual vulnerability to anxiety. This clinical study aims to develop a metacognitive task that improves existing MBCT as a new treatment that changes the function of anxiety or depression-specific neural circuits, and to explore neurological mechanisms and treatment-related factors.

This study was designed to enroll 64 participants, 32 in the NMBCT intervention and 32 in waitlist. This will allow 20% attrition and the Investigators anticipate 52 participants will complete the study. A sample size of 52 will achieve 80% power, given current effect size (cohen's d = 0.40, alpha = 0.05) estimates per aim.

Participants randomized to the NMBCT intervention or waitlist group will complete an 8-week NMBCT program conducted by a trained psychiatrist. The waitlist control group will maintain the blind for a treatment period from the baseline and then implement the NMBCT program on the NMBCT intervention group to those who agree.

Study data will be collected at 3 times for two groups: T1=1st week session (baseline); T2=8th week session; T3=6 months after baseline. All participants in the clinical study will undergo a total of two brain MRI tests within two weeks before and after visit 2 (T1, baseline) and visit 3 (T2, post-treatment, 8 weeks later).

ELIGIBILITY:
Inclusion Criteria:

* over 19 years of age
* a Beck Depression Inventory score of more than 5 but less than 20 points
* a Beck Anxiety Inventory score of more than 5 but less than 25 points
* A person who has been sufficiently explained and understood the contents of clinical trials, and maintains the ability to make a free-will decision
* Those with normal or normal corrected vision
* Those without claustrophobic symptoms
* Right-handed person
* Those who do not have a family history of psychiatric disease in the first family (parents, children, siblings)

Exclusion Criteria:

* Currently taking psychoactive drugs
* Those with a history of neurological disease, head trauma with loss of consciousness, or mental retardation (IQ <70)
* A person who currently requires hospitalization due to a serious physical illness or who has not passed 6 months since discharge
* Pregnant and lactating women
* A person who is judged to be at risk of serious suicide or violent behavior in a mental status examination
* A person who is judged to have severe symptoms or significant decline in reality testing and judgment through a mental status examination by a psychiatrist
* Foreigners
* Those who are illiterate in Korean
* Those who have previously received mindfulness-based cognitive therapy
* If the researcher judges that the researcher is unsuitable for participation in clinical trials due to other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in GMV measured with sMRI | baseline, 8 weeks after treatment
  Change in gray matter volume (GMV) in mm3 measured with structural MRI (sMRI)
Change in CT measured with sMRI | baseline, 8 weeks after treatment
  Change in cortical thickness (CT) in mm measured with structural MRI (sMRI)
Change in SA measured with sMRI | baseline, 8 weeks after treatment
  Change in surface area (SA) in mm2 measured with structural MRI (sMRI)
Change LGI measured with sMRI | baseline, 8 weeks after treatment
  Change in local gyrification index (LGI), ranged from 0 to 1, measured with structural MRI (sMRI)
Change in FA measured with DTI | baseline, 8 weeks after treatment
  Change in fractional anisotropy (FA), ranged from 0 to 1, measured with diffusion tensor imaging (DTI) and T1-weighted MR image.
Change in MD measured with DTI | baseline, 8 weeks after treatment
  Change in mean diffusivity (MD), ranged from 0 to 1, measured with diffusion tensor imaging (DTI) and T1-weighted MR image.
Change in AD measured with DTI | baseline, 8 weeks after treatment
  Change in axial diffusivity (AD), ranged from 0 to 1, measured with diffusion tensor imaging (DTI) and T1-weighted MR image.
Change in RD measured with DTI | baseline, 8 weeks after treatment
  Change in radial diffusivity (AD), ranged from 0 to 1, measured with diffusion tensor imaging (DTI) and T1-weighted MR image.
Change in FC measured with fMRI | baseline, 8 weeks after treatment
  Change in functional connectivity (FC) in resting-state functional MRI (fMRI).

SECONDARY OUTCOMES:
The changes in the Korean version of Panic Disorder Severity Scale (PDSS). | baseline, 8 week after treatment
  To assess panic symptom changes after the 8th week of treatment using the Korean version of the Panic Disorder Severity Scale (PDSS). The PDSS consists of 7 items coded on a 5-point scale (0-4). The total scores ranged from 0 to 28. The higher the total scores, the higher the panic symptom severity.
The change in the Korean version of Albany Panic and Phobia Questionnaire (APPQ) | baseline, 8 week after treatment
  To assess agoraphobia symptoms changes after the 8th week of treatment, the Korean Albany Panic and Phobia Questionnaire (APPQ) was used. The APPQ contains 27 items coded on a 9-point scale (0-8). And it can be used to assess interoceptive fear (8 items), social phobia (10 items), and agoraphobia (9 items). The higher each subscale's total score, the poorer the phobic symptom.
The change in the Korean version of the Beck Depression Inventory (BDI)-II | baseline, 8 week after treatment
  To assess depressive symptoms changes after the 8th week of treatment, the Beck Depression Inventory (BDI)-II was used. The 21 self-administered items that comprise the BDI-II were scored from a range of 0 to 3, with the maximum score being 63. The higher the total scores, the more severe the depressive symptom.
The change in the Korean version of the Beck Anxiety Inventory (BAI) | baseline, 8 week after treatment
  To assess anxiety symptoms changes after the 8th week of treatment, the Beck Anxiety Inventory (BAI) was used. The 21 self-administered items that comprise the BAI were scored from a range of 0 to 3, with the maximum score being 63. The higher the total scores, the more severe the anxiety symptom.
The change in the Korean version of the Penn State Worry Questionnaire (PSWQ) | baseline, 8 week after treatment
  To assess the frequency, intensity, and uncontrollability of pathological worry symptoms changes after the 8th week of treatment, the Penn State Worry Questionnaire (PSWQ) was used. The 16 self-administered items that comprise the PSWQ were scored from a range of 1 (not at all typical) to 5 (very typical), with the maximum score being 80. The higher the total scores, the more severe the pathological worry symptom.
The change in the Korean version of the Anxiety Sensitivity Inventory-Revised (ASI-R) | baseline, 8 week after treatment
  To assess the trait anxiety sensitivity levels changes after the 8th week of treatment, the Korean version of the Anxiety Sensitivity Inventory-Revised (ASI-R) was used. The 36-item ASI-R consists of (1) fear of respiratory symptoms, (2) publicly observable anxiety reactions, (3) cardiovascular symptoms, and (4) cognitive dyscontrol. Total scores range from 0 to 144. The higher the total scores, the higher the anxiety sensitivity levels.
The change in the Self-Compassion Scale-Short Form (SCS-SF) | baseline, 8 week after treatment
  To assess the changes in self-compassion levels after the 8th week of treatment, the Self-Compassion Scale-Short Form (SCS-SF) was used. The 12-item SCS-SF consists of self-kindness (2 items), self-judgment (2 items), common humanity (2 items), isolation subscales (2 items), mindfulness (2 items), and over-identified (2 items). Total scores range from 12 to 60. The reverse score of the negative subscale items (e.g., self-judgment, isolation, and over-identification) was used to compute total self-compassion scores. The higher the total scores, the higher the self-compassion levels.
The change in the Concise Measure of Subjective Well-Being (COMOSWB) | baseline, 8 week after treatment
  To evaluate the changes in subjective well-being levels after the 8th week of treatment, the Concise Measure of Subjective Well-Being (COMOSWB) was used. The COMOSWB consists of life satisfaction, positive affect, and negative affect. The 9-item was scored from a range of 1 (strongly disagree or never) to 7 (strongly agree or always). Total scores range from 7 to 63. The higher the total scores, the higher the subjective well-being levels.
The change in the Korean Burnout Syndrome Scale (KBOSS) | baseline, 8 week after treatment
  To evaluate the changes in burnout symptoms levels after the 8th week of treatment, the Korean Burnout Syndrome Scale (KBOSS) was used. The 12-item KBOSS consists of exhaustion (4 items), cynicism (4 items), and inefficacy (4 items). The 16-item was scored from a range of 1 (strongly disagree) to 7 (strongly agree), with the maximum score being 84. Total scores range from 12 to 84. The higher the total scores, the more severe the burn-out symptom.
The change in the Korean version of the Grit Scale | baseline, 8 week after treatment
  To evaluate the changes in grit levels after the 8th week of treatment, the Korean version of the Grit Scale was used. The 12-item of the Korean version of the Grit scale was scored from a range of 0 (strongly disagree) to 5 (strongly agree), with the maximum score being 60. The higher the total scores, the higher levels of grit.
side effects | baseline, 2 week/4 week/8 week after treatment
  To evaluate the side effects through the interview

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hyuk Lee, MD., PhD, Principal Investigator — Professor at Bundang CHA medical center

REFERENCES:
- [Background] Guendelman S, Bayer M, Prehn K, Dziobek I. Towards a mechanistic understanding of mindfulness-based stress reduction (MBSR) using an RCT neuroimaging approach: Effects on regulating own stress in social and non-social situations. Neuroimage. 2022 Jul 1;254:119059. doi: 10.1016/j.neuroimage.2022.119059. Epub 2022 Mar 5. PMID 35259523
- [Background] Yun JY, Boedhoe PSW, Vriend C, Jahanshad N, Abe Y, Ameis SH, Anticevic A, Arnold PD, Batistuzzo MC, Benedetti F, Beucke JC, Bollettini I, Bose A, Brem S, Calvo A, Cheng Y, Cho KIK, Ciullo V, Dallaspezia S, Denys D, Feusner JD, Fouche JP, Gimenez M, Gruner P, Hibar DP, Hoexter MQ, Hu H, Huyser C, Ikari K, Kathmann N, Kaufmann C, Koch K, Lazaro L, Lochner C, Marques P, Marsh R, Martinez-Zalacain I, Mataix-Cols D, Menchon JM, Minuzzi L, Morgado P, Moreira P, Nakamae T, Nakao T, Narayanaswamy JC, Nurmi EL, O'Neill J, Piacentini J, Piras F, Piras F, Reddy YCJ, Sato JR, Simpson HB, Soreni N, Soriano-Mas C, Spalletta G, Stevens MC, Szeszko PR, Tolin DF, Venkatasubramanian G, Walitza S, Wang Z, van Wingen GA, Xu J, Xu X, Zhao Q; ENIGMA-OCD working group; Thompson PM, Stein DJ, van den Heuvel OA, Kwon JS. Brain structural covariance networks in obsessive-compulsive disorder: a graph analysis from the ENIGMA Consortium. Brain. 2020 Feb 1;143(2):684-700. doi: 10.1093/brain/awaa001. PMID 32040561
- [Background] Yook K, Lee SH, Ryu M, Kim KH, Choi TK, Suh SY, Kim YW, Kim B, Kim MY, Kim MJ. Usefulness of mindfulness-based cognitive therapy for treating insomnia in patients with anxiety disorders: a pilot study. J Nerv Ment Dis. 2008 Jun;196(6):501-3. doi: 10.1097/NMD.0b013e31817762ac. PMID 18552629
- [Background] Williams LM. Precision psychiatry: a neural circuit taxonomy for depression and anxiety. Lancet Psychiatry. 2016 May;3(5):472-80. doi: 10.1016/S2215-0366(15)00579-9. Epub 2016 Apr 14. PMID 27150382
- [Background] Varghese B, Chen F, Hwang D, Palmer SL, De Castro Abreu AL, Ukimura O, Aron M, Aron M, Gill I, Duddalwar V, Pandey G. Objective risk stratification of prostate cancer using machine learning and radiomics applied to multiparametric magnetic resonance images. Sci Rep. 2019 Feb 7;9(1):1570. doi: 10.1038/s41598-018-38381-x. PMID 30733585
- [Background] Tang YY, Holzel BK, Posner MI. The neuroscience of mindfulness meditation. Nat Rev Neurosci. 2015 Apr;16(4):213-25. doi: 10.1038/nrn3916. Epub 2015 Mar 18. PMID 25783612
- [Background] Stein JL, Medland SE, Vasquez AA, Hibar DP, Senstad RE, Winkler AM, Toro R, Appel K, Bartecek R, Bergmann O, Bernard M, Brown AA, Cannon DM, Chakravarty MM, Christoforou A, Domin M, Grimm O, Hollinshead M, Holmes AJ, Homuth G, Hottenga JJ, Langan C, Lopez LM, Hansell NK, Hwang KS, Kim S, Laje G, Lee PH, Liu X, Loth E, Lourdusamy A, Mattingsdal M, Mohnke S, Maniega SM, Nho K, Nugent AC, O'Brien C, Papmeyer M, Putz B, Ramasamy A, Rasmussen J, Rijpkema M, Risacher SL, Roddey JC, Rose EJ, Ryten M, Shen L, Sprooten E, Strengman E, Teumer A, Trabzuni D, Turner J, van Eijk K, van Erp TG, van Tol MJ, Wittfeld K, Wolf C, Woudstra S, Aleman A, Alhusaini S, Almasy L, Binder EB, Brohawn DG, Cantor RM, Carless MA, Corvin A, Czisch M, Curran JE, Davies G, de Almeida MA, Delanty N, Depondt C, Duggirala R, Dyer TD, Erk S, Fagerness J, Fox PT, Freimer NB, Gill M, Goring HH, Hagler DJ, Hoehn D, Holsboer F, Hoogman M, Hosten N, Jahanshad N, Johnson MP, Kasperaviciute D, Kent JW Jr, Kochunov P, Lancaster JL, Lawrie SM, Liewald DC, Mandl R, Matarin M, Mattheisen M, Meisenzahl E, Melle I, Moses EK, Muhleisen TW, Nauck M, Nothen MM, Olvera RL, Pandolfo M, Pike GB, Puls R, Reinvang I, Renteria ME, Rietschel M, Roffman JL, Royle NA, Rujescu D, Savitz J, Schnack HG, Schnell K, Seiferth N, Smith C, Steen VM, Valdes Hernandez MC, Van den Heuvel M, van der Wee NJ, Van Haren NE, Veltman JA, Volzke H, Walker R, Westlye LT, Whelan CD, Agartz I, Boomsma DI, Cavalleri GL, Dale AM, Djurovic S, Drevets WC, Hagoort P, Hall J, Heinz A, Jack CR Jr, Foroud TM, Le Hellard S, Macciardi F, Montgomery GW, Poline JB, Porteous DJ, Sisodiya SM, Starr JM, Sussmann J, Toga AW, Veltman DJ, Walter H, Weiner MW; Alzheimer's Disease Neuroimaging Initiative; EPIGEN Consortium; IMAGEN Consortium; Saguenay Youth Study Group; Bis JC, Ikram MA, Smith AV, Gudnason V, Tzourio C, Vernooij MW, Launer LJ, DeCarli C, Seshadri S; Cohorts for Heart and Aging Research in Genomic Epidemiology Consortium; Andreassen OA, Apostolova LG, Bastin ME, Blangero J, Brunner HG, Buckner RL, Cichon S, Coppola G, de Zubicaray GI, Deary IJ, Donohoe G, de Geus EJ, Espeseth T, Fernandez G, Glahn DC, Grabe HJ, Hardy J, Hulshoff Pol HE, Jenkinson M, Kahn RS, McDonald C, McIntosh AM, McMahon FJ, McMahon KL, Meyer-Lindenberg A, Morris DW, Muller-Myhsok B, Nichols TE, Ophoff RA, Paus T, Pausova Z, Penninx BW, Potkin SG, Samann PG, Saykin AJ, Schumann G, Smoller JW, Wardlaw JM, Weale ME, Martin NG, Franke B, Wright MJ, Thompson PM; Enhancing Neuro Imaging Genetics through Meta-Analysis Consortium. Identification of common variants associated with human hippocampal and intracranial volumes. Nat Genet. 2012 Apr 15;44(5):552-61. doi: 10.1038/ng.2250. PMID 22504417
- [Background] Sun H, Chen Y, Huang Q, Lui S, Huang X, Shi Y, Xu X, Sweeney JA, Gong Q. Psychoradiologic Utility of MR Imaging for Diagnosis of Attention Deficit Hyperactivity Disorder: A Radiomics Analysis. Radiology. 2018 May;287(2):620-630. doi: 10.1148/radiol.2017170226. Epub 2017 Nov 22. PMID 29165048
- [Background] Shear MK, Bjelland I, Beesdo K, Gloster AT, Wittchen HU. Supplementary dimensional assessment in anxiety disorders. Int J Methods Psychiatr Res. 2007;16 Suppl 1(Suppl 1):S52-64. doi: 10.1002/mpr.215. PMID 17623395
- [Background] Roy-Byrne PP, Craske MG, Stein MB. Panic disorder. Lancet. 2006 Sep 16;368(9540):1023-32. doi: 10.1016/S0140-6736(06)69418-X. PMID 16980119
- [Background] Park YW, Choi D, Lee J, Ahn SS, Lee SK, Lee SH, Bang M. Differentiating patients with schizophrenia from healthy controls by hippocampal subfields using radiomics. Schizophr Res. 2020 Sep;223:337-344. doi: 10.1016/j.schres.2020.09.009. Epub 2020 Sep 26. PMID 32988740
- [Background] Park JE, Kim HS. Radiomics as a Quantitative Imaging Biomarker: Practical Considerations and the Current Standpoint in Neuro-oncologic Studies. Nucl Med Mol Imaging. 2018 Apr;52(2):99-108. doi: 10.1007/s13139-017-0512-7. Epub 2018 Feb 1. PMID 29662558
- [Background] Liang S, Ma A, Yang S, Wang Y, Ma Q. A Review of Matched-pairs Feature Selection Methods for Gene Expression Data Analysis. Comput Struct Biotechnol J. 2018 Feb 25;16:88-97. doi: 10.1016/j.csbj.2018.02.005. eCollection 2018. PMID 30275937
- [Background] Klauke B, Deckert J, Reif A, Pauli P, Domschke K. Life events in panic disorder-an update on "candidate stressors". Depress Anxiety. 2010 Aug;27(8):716-30. doi: 10.1002/da.20667. PMID 20112245
- [Background] Kim YW, Lee SH, Choi TK, Suh SY, Kim B, Kim CM, Cho SJ, Kim MJ, Yook K, Ryu M, Song SK, Yook KH. Effectiveness of mindfulness-based cognitive therapy as an adjuvant to pharmacotherapy in patients with panic disorder or generalized anxiety disorder. Depress Anxiety. 2009;26(7):601-6. doi: 10.1002/da.20552. PMID 19242985
- [Background] Kim MK, Kim B, Kiu Choi T, Lee SH. White matter correlates of anxiety sensitivity in panic disorder. J Affect Disord. 2017 Jan 1;207:148-156. doi: 10.1016/j.jad.2016.08.043. Epub 2016 Oct 3. PMID 27721189
- [Background] Insel TR, Cuthbert BN. Medicine. Brain disorders? Precisely. Science. 2015 May 1;348(6234):499-500. doi: 10.1126/science.aab2358. No abstract available. PMID 25931539
- [Background] Harrison BJ, Fullana MA, Soriano-Mas C, Via E, Pujol J, Martinez-Zalacain I, Tinoco-Gonzalez D, Davey CG, Lopez-Sola M, Perez Sola V, Menchon JM, Cardoner N. A neural mediator of human anxiety sensitivity. Hum Brain Mapp. 2015 Oct;36(10):3950-8. doi: 10.1002/hbm.22889. Epub 2015 Jul 6. PMID 26147233
- [Background] Hamilton SP, Slager SL, De Leon AB, Heiman GA, Klein DF, Hodge SE, Weissman MM, Fyer AJ, Knowles JA. Evidence for genetic linkage between a polymorphism in the adenosine 2A receptor and panic disorder. Neuropsychopharmacology. 2004 Mar;29(3):558-65. doi: 10.1038/sj.npp.1300311. PMID 14666117
- [Background] Fraguas D, Diaz-Caneja CM, State MW, O'Donovan MC, Gur RE, Arango C. Mental disorders of known aetiology and precision medicine in psychiatry: a promising but neglected alliance. Psychol Med. 2017 Jan;47(2):193-197. doi: 10.1017/S0033291716001355. Epub 2016 Jun 23. PMID 27334937
- [Background] Dow MG, Kenardy JA, Johnston DW, Newman MG, Taylor CB, Thomson A. Prognostic indices with brief and standard CBT for panic disorder: I. Predictors of outcome. Psychol Med. 2007 Oct;37(10):1493-502. doi: 10.1017/S0033291707000670. Epub 2007 May 10. PMID 17493294
- [Background] Black DW, Wesner RB, Gabel J, Bowers W, Monahan P. Predictors of short-term treatment response in 66 patients with panic disorder. J Affect Disord. 1994 Apr;30(4):233-41. doi: 10.1016/0165-0327(94)90131-7. PMID 8014323
- [Background] Angst J, Vollrath M. The natural history of anxiety disorders. Acta Psychiatr Scand. 1991 Nov;84(5):446-52. doi: 10.1111/j.1600-0447.1991.tb03176.x. PMID 1776498